CLINICAL TRIAL: NCT05523206
Title: A Natural History Study of Biomarkers and Clinical Outcomes in Mucopolysaccharidosis Type IIIA (MPS IIIA)
Brief Title: A Natural History Study of Biomarkers and Clinical Outcomes in Mucopolysaccharidosis Type IIIA (MPS IIIA; Sanfilippo Syndrome)
Status: Completed | Type: Observational
Sponsor: Sanguine Biosciences (Industry)
Collaborators: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SAN-08252
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Mucopolysaccharidosis III-A
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with MPS IIIA
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This protocol is a decentralized, single cohort, natural history and biomarker study enrolling up to 20 participants with MPS IIIA (Sanfilippo syndrome). At least 10 participants (~50%) must be less than four years old at the time of the Parent/LAR consent. The study will have a screening process and 7 study visits, e.g. home visits, that will consist of serum collection and completion of a remote assessment of the Vineland Adaptive Behavior Scales 3rd Edition (Vineland-3)

MPS IIIA remains a devastating disease with a high unmet medical need. There is currently a limited number of available data to adequately characterize the progression of the disease. Analysis of blood biospecimens and adaptive behavior in this study will help researchers better understand the clinical progression of MPS IIIA. A better understanding of disease progression may assist in developing novel therapies for rare genetic disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age of enrollment is as follows:

  1. All participants must be between 4 months and < 14 years at time of consent
  2. At least 10 participants (ie, approx. 50% of expected total population) must be between 4 months old and < 4 years old at the time of consent
* The participant has a confirmed diagnosis of Mucopolysaccharidosis Type IIIA (MPS IIIA) (i.e., Sanfilippo syndrome) based on at least 2 out of the 3 following criteria:

  1. Documented reduced N-sulphoglucosamine sulphohydrolase (SGSH) activity in plasma, white blood cells, and/or skin fibroblasts consistent with MPS IIIA (10% or less of the lower limit of the normal range based on the testing laboratory)
  2. Documented likely pathogenic variant of the SGSH gene
  3. Documented elevated heparan sulfate levels in urine and/or blood Participants and their families are willing to complete 7 blood draws and 7 Vineland-3 collections

Exclusion Criteria:

* Known history of HIV, hepatitis, or other infectious diseases
* Taken an investigational product in the last 30 days
* Experienced excess blood loss, including blood donation, defined as 80 mL in the last month or 160 mL in the previous two months
* Undergone an MPS IIIA gene therapy at any time unless prior Sponsor or designee's approval has been received
* Documented loss of activity of sulfatases other than N-sulphoglucosamine sulphohydrolase (SGSH), indicating multiple sulfatase deficiency
* Known genetic or acquired disorder associated with developmental delay, seizures or other significant CNS dysfunction that would be expected to confound the clinical or biomarker assessments

Ages: 4 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participant eligibility is based on age and on a confirmed diagnosis of Mucopolysaccharidosis Type IIIA (Sanfilippo syndrome).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline of adaptive behavior as measured by remote administration of the Vineland-3 Adaptive Behavior Scales (Vineland-3) | 96 weeks
Change from baseline in levels of blood-based biomarkers in serum | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Houman Hemmati, MD, Principal Investigator — Sanguine Biosciences, Inc.
Locations (1):
- Sanguine Biosciences, Inc., Woburn, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No